CLINICAL TRIAL: NCT02729792
Title: Canadian rTMS Treatment and Biomarker Network in Depression Trial
Acronym: CARTBIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University Health Network, Toronto (Other); University of British Columbia (Other); Brain Canada (Other)
Responsible Party: Principal Investigator, Daniel Blumberger, Medical Head and Co-Director, Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 052-2015
Record Dates: First submitted 2016-03-29; First posted 2016-04-06 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Depression
Keywords: depression; treatment resistance; biomarkers; repetitive transcranial magnetic stimulation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single site rTMS (Experimental): Each treatment session will consist of:
  1200 pulses of iTBS over a posterior target location followed by a 60 minute interval, then 1200 pulses of iTBS over an anterior target location.
  Interventions: Device: rTMS
- Dual site rTMS (Active Comparator): Each treatment session will consist of:
  600 pulses of iTBS over the posterior target, followed immediately by 600 pulses of iTBS over the anterior target location followed by a 60 minute interval, then 600 pulses of iTBS over the posterior target, followed immediately by 600 pulses of iTBS over the anterior target location.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — intermittent theta burst stimulation (iTBS)

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) is an emerging treatment for medically refractory major depressive disorder (MDD). rTMS involves direct stimulation of cortical neurons using externally applied, powerful, focused magnetic field pulses. Dozens of studies and several meta-analyses over the last 15 years have shown that rTMS of the dorsolateral prefrontal cortex (DLPFC) produces statistically significant improvements in MDD, even when medications have failed. However, other possible targets may also yield improvement in symptoms.

In an attempt to enhance the therapeutic efficacy of current interventions for TRD, attention has turned to identifying domain-specific biomarkers in hopes of ultimately individualizing and predicting treatment response. Unfortunately, the precise nature of this relationship is less than clear, as reflected by the fact that even now there are no established biomarkers that are used routinely in clinical practice to aid in diagnosis. This study also seeks to examine a comprehensive suite of biomarker measurements (MRI, neurophysiology, and genomics/proteomics) before and after rTMS treatment.

DETAILED DESCRIPTION:
rTMS is a Health-Canada- and FDA-approved treatment for treatment-resistant depression (TRD), using focused magnetic field pulses to stimulate brain regions involved in emotion regulation, safely and non-invasively. Though rTMS is often effective where medications or therapy fail, it requires a series of lengthy (~30-40 min) treatment sessions. A new form of rTMS called theta burst stimulation (TBS) has been shown to have greater effects on neural activity than conventional stimulation, despite requiring as little as 40 s of stimulation. The purpose of this study is to assess the efficacy and tolerability of an accelerated TBS protocol, administered 2 times a day in patients with TRD. In addition, the investigators aim to identify candidate biomarkers from a multimodal suite of neuroimaging, neurophysiologic and molecular measures that are predictors and correlates of response to rTMS treatment.

ELIGIBILITY:
Inclusion Criteria:

1. are outpatients
2. are voluntary and competent to consent to treatment
3. have a Mini-International Neuropsychiatric Interview (MINI) confirmed diagnosis of MDD, single or recurrent
4. are between the ages of 18 and 59
5. have failed to achieve a clinical response to an adequate dose of an antidepressant based on an Antidepressant Treatment History Form (ATHF) score for that antidepressant trial of > 3 in the current episode 105,106 OR have been unable to tolerate at least 2 separate trials of antidepressants of inadequate dose and duration (ATHF score of 1 or 2 on those 2 separate antidepressants)
6. have a score > 18 on the HRSD-17 item
7. have had no increase or initiation of any psychotropic medication in the 4 weeks prior to screening
8. able to adhere to the treatment schedule
9. Pass the TMS adult safety screening (TASS) questionnaire
10. have normal thyroid functioning based on pre-study blood work.

Exclusion Criteria:

1. have a Mini-International Neuropsychiatric Interview (MINI) confirmed diagnosis of substance dependence or abuse within the last 3 months
2. have a concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump
3. have active suicidal intent
4. are pregnant
5. have a lifetime Mini-International Neuropsychiatric Interview (MINI) diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms
6. have a MINI diagnosis of obsessive compulsive disorder, post-traumatic stress disorder (current or within the last year), anxiety disorder (generalized anxiety disorder, social anxiety disorder, panic disorder), or dysthymia, assessed by a study investigator to be primary and causing greater impairment than MDD
7. have a diagnosis of any personality disorder, and assessed by a study investigator to be primary and causing greater impairment than MDD
8. have failed a course of ECT in the current episode or previous episode
9. have received rTMS for any previous indication due to the potential compromise of subject blinding
10. have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of seizure except those therapeutically induced by ECT or a febrile seizure of infancy, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than 5 minutes
11. have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
12. if participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study
13. clinically significant laboratory abnormality, in the opinion of the one of the principal investigators or study physicians
14. currently take more than lorazepam 2 mg daily (or equivalent) or any dose of an anticonvulsant due to the potential to limit rTMS efficacy
15. non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 212 (Actual)
Dates: Start 2016-03; Primary Completion 2018-02-23 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
17-item Hamilton Rating Scale for Depression (HRSD-17) Change | 10 days
  Change from baseline to 10 days

SECONDARY OUTCOMES:
17-item Hamilton Rating Scale for Depression (HRSD-17) Change | 30 days
  Change from baseline to 30 days

OTHER OUTCOMES:
Beck Depression Inventory-II Change | 10 days
  Change from baseline to 10 days
Quick Inventory of Depressive Symptoms Change | 10 days
  Change from baseline to 10 days
17-item Hamilton Rating Scale for Depression (HRSD-17) Remission | 10 days
  Remission rates defined as a HRSD-17 < 8 at 10 days
Beck Depression Inventory-II | 30 days
  Change from baseline to 30 days
Quick Inventory of Depressive Symptoms Change | 30 Days
  Change from baseline to 30 days
17-item Hamilton Rating Scale for Depression (HRSD-17) Remission | 30 days
  Remission rates defined as a HRSD-17 < 8 at 30 days
17-item Hamilton Rating Scale for Depression (HRSD-17) Response | 10 days
  Response rates defined as a HRSD-17 decrease > 50% at 10 days
17-item Hamilton Rating Scale for Depression (HRSD-17) Response | 30 days
  Response rates defined as a HRSD-17 decrease > 50% at 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M. Blumberger, MD, MSc, Principal Investigator — CAMH
Locations (3):
- Canada (3):
  - Non-Invasive Neurostimulation Therapies Centre, University of British Columbia, Vancouver, British Columbia
  - Toronto Western Hospital, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen X, Blumberger DM, Yan CG, Downar J, Vila-Rodriguez F, Daskalakis ZJ, Kaster TS. Crosswalk between HRSD and MADRS outcomes for rTMS in patients with depression. BMJ Ment Health. 2025 Mar 28;28(1):e301451. doi: 10.1136/bmjment-2024-301451. PMID 40154967
- [Derived] Zapf L, Kaster TS, Vila-Rodriguez F, Daskalakis ZJ, Downar J, Blumberger DM. The effect of once-daily vs. twice-daily intermittent theta burst stimulation on suicidal ideation in treatment-resistant depression. Eur Arch Psychiatry Clin Neurosci. 2025 Sep;275(6):1787-1798. doi: 10.1007/s00406-024-01929-2. Epub 2024 Nov 15. PMID 39545967
- [Derived] Kaster TS, Downar J, Vila-Rodriguez F, Baribeau DA, Thorpe KE, Daskalakis ZJ, Blumberger DM. Differential symptom cluster responses to repetitive transcranial magnetic stimulation treatment in depression. EClinicalMedicine. 2022 Dec 2;55:101765. doi: 10.1016/j.eclinm.2022.101765. eCollection 2023 Jan. PMID 36483268
- [Derived] Blumberger DM, Vila-Rodriguez F, Wang W, Knyahnytska Y, Butterfield M, Noda Y, Yariv S, Isserles M, Voineskos D, Ainsworth NJ, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. A randomized sham controlled comparison of once vs twice-daily intermittent theta burst stimulation in depression: A Canadian rTMS treatment and biomarker network in depression (CARTBIND) study. Brain Stimul. 2021 Nov-Dec;14(6):1447-1455. doi: 10.1016/j.brs.2021.09.003. Epub 2021 Sep 21. PMID 34560319
- See also: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — http://www.camh.ca/en/research